CLINICAL TRIAL: NCT04168125
Title: Use of Tilapia Skin for Palate Repair and Protection After Graft Removal
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Gustavo Gonçalves do Prado Manfredi, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ceap
Record Dates: First submitted 2019-09-27; First posted 2019-11-19 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Pain, Postoperative; Palate; Wound; Cicatrization
MeSH Terms: conditions — Pain, Postoperative; Wounds and Injuries; Cicatrix

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tilapia skin (Experimental): Procedure/Surgery: Free gingival graft harvesting from hard palate. After gingival graft harvesting from hard palate, it will be placed a tilapia skin as an occlusive biological dressing for palatal wound healing.
  Device: Tilapia skin. A xenogeneic collagen dressing will be placed over palate wound and stabilized with sutures during the healing process.
  Interventions: Device: Tilapia skin
- Surgical Wound Dressing (Active Comparator): Procedure/Surgery: Free gingival graft harvesting from hard palate. After gingival graft harvesting from hard palate, it will be placed a surgical wound dressing as a mechanical protection during palatal wound healing.
  Device: Surgical wound dressing A surgical wound dressing will be placed over palate wound during the healing process to provide mechanical protection.
  Interventions: Device: Surgical Wound Dressing

INTERVENTIONS:
Device: Tilapia skin — Application tilapia skin as an occlusive biological dressing for palatal wound healing after free gingival graft harvesting.
  Arms: Tilapia skin
Device: Surgical Wound Dressing — Application surgical wound dressing as an occlusive biological dressing for palatal wound healing after free gingival graft harvesting.
  Arms: Surgical Wound Dressing

SUMMARY:
Randomised Clinical Study to evaluate the efficacy of tilapia skin as an occlusive biological dressing on palatal wound healing after free gingival graft harvesting.

DETAILED DESCRIPTION:
Autogenous grafts are currently considered the gold standard in regenerative and reconstructive procedures. However, these procedures require a second surgical site to provide the tissue graft. In autogenous gingival grafts, the area commonly selected for graft harvesting is the palate, which is linked to great discomfort and morbidity for the patient. In order to overcome these limitations, xenogeneic and alloplastic materials have been tested as tissue substitutes, but their results are still considerably inferior when compared to autogenous grafts. Faced with this superiority, another approach to favor the use of autogenous grafting is to develop materials that provide greater postoperative comfort and patient safety. Since the main complaint arising from the technique is related to pain resulting from the remaining surgical wound on the palate, it is interesting to look for mechanisms to reduce this sensitivity and accelerate the healing process. For this, the use of tilapia skin as a postoperative dressing seems to be a good alternative. Thus, the purpose of this study is to evaluate the use of tilapia skin, with the intention of accelerating the palate healing process, and to serve as a protector barrier during the healing process. Patients treated according to two techniques for palate protection after autogenous gingival graft harvesting will be evaluated: C- use of surgical cement and T- use of tilapia skin. Will be selected 60 patients of both sexes,> 18 years old, requiring the removal of the palate graft for periodontal surgery. At the time of graft removal, palate thickness and graft dimensions will be measured. After 7, 14 and 30 days, the patient's discomfort and the difficulty in chewing and speaking will be recorded through a visual analog scale, the consumption of analgesic, and the dimensions of the surgical wound on the palate. For statistical analysis, two-way ANOVA will be performed and t-test paired on the obtained results.

ELIGIBILITY:
Inclusion Criteria:

* Patients need periodontal or peri-implant surgical procedures requiring palate gingival graft

Exclusion Criteria:

* Patients with an infectious condition that compromises the procedures
* Users of drugs that can act on periodontal tissues or the healing process
* Pregnant
* Smokers
* Diabetes
* Irradiated

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
Self-reported pain perception evaluated by a visual analog scale | 14 days after the surgery
  Patient's self-reported pain perception will be evaluated using a visual analog scale with a score ranging from 0 (no pain) to 10 (unbearable pain).

SECONDARY OUTCOMES:
Self-reported discomfort evaluated by a visual analog scale | 14 days after the surgery
  Patient's self-reported discomfort will be evaluated using a visual analog scale with a score ranging from 0 (no discomfort) to 2 (high discomfort).
Self-reported trouble with speech evaluated by a visual analog scale | 14 days after the surgery
  Patient's self-reported trouble with speech will be evaluated using a visual analog scale with a score ranging from 0 (no trouble) to 2 (high trouble).
Self-reported trouble with eating evaluated by a visual analog scale | 14 days after the surgery
  Patient's self-reported trouble with eating will be evaluated using a visual analog scale with a score ranging from 0 (no trouble) to 2 (high trouble).
Comparison of the palate healing process evaluated through linear measurements (millimiter) | 30 days after the surgery
  Pictures will be taken immediately after the gingival graft harvesting and compared with post-operativa pictures through the use of linear measurements at Image J.
Number of analgesic pills taken after surgery | 14 days after the surgery
  Evaluate the patient's perception of postoperative pain and discomfort by counting the number of analgesic pills taken after the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana CP Sant'Ana, PhD, Study Director — Bauru School of Dentistry - University of Sao Paulo
Locations (1):
- Bauru School of Dentistry, Bauru, Brazil, Brazil

IPD SHARING:
Plan to Share IPD: No